CLINICAL TRIAL: NCT04219033
Title: Correlation Between Postoperative Cognitive Function and EEG Parameters in Elderly Patients Undergoing Non-cardiac Major Surgery : Multi-center, Prospective, Observational Study
Brief Title: Postoperative Cognitive Function and EEG
Acronym: POEM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Zhihong LU, professor, Air Force Military Medical University, China
Other Study IDs: XJH-A-20190726
Record Dates: First submitted 2019-12-31; First posted 2020-01-06 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-10

CONDITIONS: Aging; Postoperative Cognitive Dysfunction; EEG With Periodic Abnormalities
Keywords: noncardiac surgery; elderly patients; postoperative cognitive dysfunction; Electroencephalogram
MeSH Terms: conditions — Postoperative Cognitive Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- with postoperative cognitive dysfunction
  Interventions: Other: EEG(Electroencephalogram) change
- without postoperative dysfunction
  Interventions: Other: EEG(Electroencephalogram) change

INTERVENTIONS:
Other: EEG(Electroencephalogram) change — patients are found to have characteristic EEG change

SUMMARY:
In the elderly patients undergoing elective non-cardiac major surgery, the differences of EEG parameters between those with and without postoperative cognitive dysfunction were observed to determine the characteristic changes of EEG parameters related to postoperative cognitive dysfunction

ELIGIBILITY:
Inclusion Criteria:

1. aged 65 and above
2. non-cardiac surgery under general anesthesia;
3. American Society of Anesthesiology(ASA) classification I- II
4. Patients aged 18-40 years old are set as background

Exclusion Criteria:

1. patients with central nervous system diseases and mental diseases
2. preoperative minimal mental status examination(MMSE) score<24;
3. ASA status III or higher

3) those who have received less than 5 years of education since entering primary school; 4) history of sedatives or antidepressants use; 5) existed or anticipated alcohol or drug abuse(over 40°c and over 100ml per day for the past 3 months); 6) history of surgery within the previous year; 7) those with severe visual or hearing impairment; 8) those participated in other clinical studies within last 3 months;

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: 1150 cases in the elderly group and 100 cases in the adult background group
Sampling Method: Probability Sample
Enrollment: 1250 (Estimated)
Dates: Start 2020-05-05 (Actual); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
The difference of delta wave miss rate between patients with or without cognitive dysfunction by 1 day after surgery | from end of surgery to 1 day after surgery
  The difference (OR) between the miss rate of delta wave in patients with and without cognitive function change 1 day after operation.
The difference of spindle miss rate between patients with or without cognitive dysfunction by 1day after surgery | from end of surgery to 1 day after surgery
  The difference (OR) between the miss rate of spindle in patients with and without cognitive function change 1 day after operation.

SECONDARY OUTCOMES:
The difference of delta wave miss rate between patients with or without cognitive dysfunction by 3 days after surgery | from end of surgery to 3 day after surgery
The difference of spindle miss rate between patients with or without cognitive dysfunction by 3 days after surgery | from end of surgery to 3 days after surgery
The difference of burst suppression rate between patients with or without cognitive dysfunction by 3 days after surgery | from end of surgery to 3 days after surgery
correlation of delta wave miss rate and incidence of postoperative cognitive dysfunction by 1 day after surgery | from end of surgery to 1 day after surgery
correlation of delta wave miss rate and incidence of postoperative cognitive dysfunction by 3 days after surgery | from end of surgery to 3 days after surgery
correlation of spindle miss rate and incidence of postoperative cognitive dysfunction by 1d after surgery | from end of surgery to 1d after surgery
correlation of spindle miss rate and incidence of postoperative cognitive dysfunction by 3 days after surgery | from end of surgery to 3 days after surgery
correlation of burst suppression rate and incidence of postoperative cognitive dysfunction by 1 day after surgery | from end of surgery to 1 day after surgery
correlation of burst suppression rate and incidence of postoperative cognitive dysfunction by 3 days after surgery | from end of surgery to 3 days after surgery
correlation of burst suppression rate and incidence of death by 30 days after surgery | from end of surgery to 30 days after surgery
correlation of delta wave miss rate and incidence of death by 30 days after surgery | from end of surgery to 30 days after surgery
correlation of spindle miss rate and incidence of death by 30 days after surgery | from end of surgery to 30 days after surgery

CONTACTS AND LOCATIONS:
Locations (18):
- China (18):
  - Suzhou First People's Hospital, Suzhou, Jiangsu
  - The First Affiliated Hospital Nanchang University, Nanchang, Jiangxi
  - General Hospital of Northern Theater Command, Shenyang, Liaoning
  - General Hospital of Ningxia Medical University, Yinchuan, Ningxia
  - Qinhai Provincial People's Hospital, Xining, Qinghai
  - The Second Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - First Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Second Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Shanxi Bethune Hospital, Taiyuan, Shanxi
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - China-Japan Friendship Hospital, Beijing
  - Xinqiao Hospital of Army Medical University, Chongqing
  - People's Hospital of Jiangsu, Nanjing
  - Weinan Central Hospital, Weinan
  - Zhongnan Hospital of Wuhan University, Wuhan
  - People's Hospital of Zhanjiang, Zhanjiang
  - People's Hospital of Zhengzhou University, Zhengzhou
  - Traditional Chinese Medicine Hospital of Henan, Zhengzhou

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Vutskits L, Xie Z. Lasting impact of general anaesthesia on the brain: mechanisms and relevance. Nat Rev Neurosci. 2016 Oct 18;17(11):705-717. doi: 10.1038/nrn.2016.128. PMID 27752068
- [Result] Monk TG, Weldon BC, Garvan CW, Dede DE, van der Aa MT, Heilman KM, Gravenstein JS. Predictors of cognitive dysfunction after major noncardiac surgery. Anesthesiology. 2008 Jan;108(1):18-30. doi: 10.1097/01.anes.0000296071.19434.1e. PMID 18156878
- [Result] Abildstrom H, Rasmussen LS, Rentowl P, Hanning CD, Rasmussen H, Kristensen PA, Moller JT. Cognitive dysfunction 1-2 years after non-cardiac surgery in the elderly. ISPOCD group. International Study of Post-Operative Cognitive Dysfunction. Acta Anaesthesiol Scand. 2000 Nov;44(10):1246-51. doi: 10.1034/j.1399-6576.2000.441010.x. PMID 11065205